CLINICAL TRIAL: NCT05830747
Title: Three-dimensional Facial Swelling Evaluation of Pre-operative Single-dose of Prednisone in Third Molar Surgery: a Split-mouth Randomized Controlled Trial
Brief Title: Effect of Pre-emptive Dose of Prednisone Versus Placebo in Impacted Third Molar Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Magna Graecia (Other)
Responsible Party: Principal Investigator, Amerigo Giudice, Professor, University Magna Graecia
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 465/2020
Record Dates: First submitted 2023-03-27; First posted 2023-04-26 (Actual); Last update posted 2023-04-26 (Actual); Status verified 2023-04

CONDITIONS: Facial Swelling; Tooth Position Anomalies; Tooth, Impacted; Tooth Extraction Status Nos; Tooth Avulsion
Keywords: third molar surgery; facial swelling; 3D facial swelling evaluation; tooth impacted; prednisone drug administration; corticosteroids administration
MeSH Terms: conditions — Tooth, Impacted; Tooth Avulsion | interventions — Prednisone

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Prednisone group (PG) (Experimental): Patients receiving a preoperative administration of prednisone 25 mg/os.
  Interventions: Drug: Prednisone
- Control group (CG) (Placebo Comparator): Patients receiving a preoperative administration of Placebo.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Prednisone — Pre-operative drug administration before third molar surgery
  Arms: Prednisone group (PG)
Drug: Placebo — Pre-operative Placebo administration before third molar surgery
  Arms: Control group (CG)

SUMMARY:
The present study proposes to compare the effect of a single preoperative dose of prednisone versus placebo in terms of facial swelling, trismus and pain after surgical removal of the mandibular third molar (M3M) in a split-mouth randomized controlled clinical trial.

DETAILED DESCRIPTION:
This study aims to compare the effect of a single preoperative dose of prednisone versus placebo in terms of facial swelling, trismus, and pain after surgical removal of M3M in a split-mouth randomized controlled clinical trial. Facial swelling will be evaluated using an innovative three-dimensional digital technique.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 to 32 years who required both M3M extractions were recruited
* Good health status
* Indication to surgical extraction of both M3M
* Complete root formation
* Surgical risk level classified as "Conventional" or "Moderate" according to Daugela et al. classification

Exclusion Criteria:

* Person under the age of 18 or over 32
* Allergy or contraindications to administration of corticosteroids
* Acute infection in any of the teeth to be extracted
* Patients with chronic liver disease, diabetes, immune system dysfunction, or haematological disease
* Pregnancy or breastfeeding
* History of treatment with antiresorptive drugs
* Chronic kidney disease
* History of systemic corticosteroid therapy in the past 4 weeks

Ages: 18 Years to 32 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2022-10-25 (Actual); Study Completion 2022-12-10 (Actual)

PRIMARY OUTCOMES:
Change in facial swelling | Change from baseline (before surgery) at 2 day after surgery and at 7 days after surgery
  To compare the effectiveness of prednisone/os versus placebo in reducing facial swelling using qualitative three-dimensional analysis (measured by colorimetric variation given by the overlapping volumes) .
Change in facial swelling | Change from baseline (before surgery) at 2 day after surgery and at 7 days after surgery
  To compare the effectiveness of prednisone/os versus placebo in reducing facial swelling using quantitative three-dimensional analysis (differences are measured in cm3).

SECONDARY OUTCOMES:
Change in trismus | Change from baseline (before surgery) at 2 day after surgery and at 7 days after surgery
  To assess the effects of prednisone/os administration on trismus (measured in cm)
Change in pain with Visual analogue scale (VAS) | Change from baseline (before surgery) at 2 day after surgery and at 7 days after surgery
  To assess the effects of prednisone/os administration on pain (measured by VAS-score from 0 to 10 point, with 10 as the worst outcome)

CONTACTS AND LOCATIONS:
Overall Officials: Alessandro Antonelli, PhDs, DDS, Principal Investigator — Magna Graecia University of Catanzaro
Locations (1):
- Magna Graecia University of Catanzaro, Catanzaro, CZ, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Cankaya AB, Akcay C, Kahraman N, Koseoglu BG. Oral surgical procedures under local anaesthesia in day surgery. BMC Oral Health. 2018 Oct 30;18(1):179. doi: 10.1186/s12903-018-0648-6. PMID 30376855
- [Result] Sifuentes-Cervantes JS, Carrillo-Morales F, Castro-Nunez J, Cunningham LL, Van Sickels JE. Third molar surgery: Past, present, and the future. Oral Surg Oral Med Oral Pathol Oral Radiol. 2021 Nov;132(5):523-531. doi: 10.1016/j.oooo.2021.03.004. Epub 2021 Mar 14. PMID 34030996
- [Result] Sainz de Baranda B, Silvestre FJ, Silvestre-Rangil J. Relationship Between Surgical Difficulty of Third Molar Extraction Under Local Anesthesia and the Postoperative Evolution of Clinical and Blood Parameters. J Oral Maxillofac Surg. 2019 Jul;77(7):1337-1345. doi: 10.1016/j.joms.2019.02.020. Epub 2019 Feb 20. PMID 30878593
- [Result] Yamalik K, Bozkaya S. The predictivity of mandibular third molar position as a risk indicator for pericoronitis. Clin Oral Investig. 2008 Mar;12(1):9-14. doi: 10.1007/s00784-007-0131-2. Epub 2007 Jul 10. PMID 17619915
- [Result] Yoo JH, Yeom HG, Shin W, Yun JP, Lee JH, Jeong SH, Lim HJ, Lee J, Kim BC. Deep learning based prediction of extraction difficulty for mandibular third molars. Sci Rep. 2021 Jan 21;11(1):1954. doi: 10.1038/s41598-021-81449-4. PMID 33479379
- [Result] Acham S, Klampfl A, Truschnegg A, Kirmeier R, Sandner-Kiesling A, Jakse N. Beneficial effect of methylprednisolone after mandibular third molar surgery: a randomized, double-blind, placebo-controlled split-mouth trial. Clin Oral Investig. 2013 Sep;17(7):1693-700. doi: 10.1007/s00784-012-0867-1. Epub 2012 Oct 30. PMID 23108628
- [Result] Herrera-Briones FJ, Prados Sanchez E, Reyes Botella C, Vallecillo Capilla M. Update on the use of corticosteroids in third molar surgery: systematic review of the literature. Oral Surg Oral Med Oral Pathol Oral Radiol. 2013 Nov;116(5):e342-51. doi: 10.1016/j.oooo.2012.02.027. Epub 2012 Aug 17. PMID 22902498
- [Result] Ngeow WC, Lim D. Do Corticosteroids Still Have a Role in the Management of Third Molar Surgery? Adv Ther. 2016 Jul;33(7):1105-39. doi: 10.1007/s12325-016-0357-y. Epub 2016 Jun 10. PMID 27287853
- [Result] Tiigimae-Saar J, Leibur E, Tamme T. The effect of prednisolone on reduction of complaints after impacted third molar removal. Stomatologija. 2010;12(1):17-22. PMID 20440092
- [Result] Kaewkumnert S, Phithaksinsuk K, Changpoo C, Nochit N, Muensaiyat Y, Wilaipornsawai S, Piriyaphokai U, Powcharoen W. Comparison of intraosseous and submucosal dexamethasone injection in mandibular third molar surgery: a split-mouth randomized clinical trial. Int J Oral Maxillofac Surg. 2020 Apr;49(4):529-535. doi: 10.1016/j.ijom.2019.10.006. Epub 2019 Oct 25. PMID 31668666
- [Result] Juodzbalys G, Daugela P. Mandibular third molar impaction: review of literature and a proposal of a classification. J Oral Maxillofac Res. 2013 Jul 1;4(2):e1. doi: 10.5037/jomr.2013.4201. PMID 24422029
- [Result] Lau AAL, De Silva RK, Thomson M, De Silva H, Tong D. Third Molar Surgery Outcomes: A Randomized Clinical Trial Comparing Submucosal and Intravenous Dexamethasone. J Oral Maxillofac Surg. 2021 Feb;79(2):295-304. doi: 10.1016/j.joms.2020.09.020. Epub 2020 Sep 17. PMID 33058774
- [Derived] Antonelli A, Barone S, Bennardo F, Giudice A. Three-dimensional facial swelling evaluation of pre-operative single-dose of prednisone in third molar surgery: a split-mouth randomized controlled trial. BMC Oral Health. 2023 Aug 31;23(1):614. doi: 10.1186/s12903-023-03334-y. PMID 37653378